CLINICAL TRIAL: NCT01223365
Title: A 12-Month, Open-Label Study to Evaluate the Long-Term Safety of Hydrocodone Bitartrate Extended-Release Tablets (CEP-33237) at 15 to 90 mg Every 12 Hours in Patients Who Require Opioid Treatment for an Extended Period of Time
Brief Title: Study to Evaluate the Long-Term Safety of Hydrocodone Bitartrate Extended-Release Tablets (CEP-33237) in Patients Who Require Opioid Treatment for an Extended Period of Time
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C33237/3080
Record Dates: First submitted 2010-10-15; First posted 2010-10-19 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Chronic Pain
Keywords: moderate to severe pain; diabetic peripheral neuropathy; postherpetic neuralgia; traumatic injury; complex regional pain syndrome; back pain; neck pain; osteoarthritis; rheumatoid arthritis
MeSH Terms: conditions — Chronic Pain; Neuralgia, Postherpetic; Wounds and Injuries; Complex Regional Pain Syndromes; Back Pain; Neck Pain; Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydrocodone ER (Experimental): Participants were titrated (or re-titrated for roll-over participants) at escalating dosages of extended-release hydrocodone tablets at dosages of 15, 30, 45, 60, or 90 mg orally every 12 hours until deemed successful for managing their pain during the open-label titration period. Once a successful dose was identified, participants entered the 52 week open-label treatment period in which hydrocodone ER was administered at the successful dose (15, 30, 45, 60, or 90 mg) every 12 hours.
  Interventions: Drug: Hydrocodone ER

INTERVENTIONS:
Drug: Hydrocodone ER — Hydrocodone bitartrate extended-release tablets were administered at doses of 15, 30, 45, 60, and 90 mg orally every 12 hours. During the open-label titration period, doses were adjusted until a stable pain control was achieved. In general, the dose of hydrocodone extended release tablets could be adjusted for efficacy or tolerability, as necessary, at any time during the open-label treatment period; however, participants were required to visit the study center before increasing the dose of study drug.
  Other Names: CEP-33237; Hydrocodone bitartrate extended-release

SUMMARY:
The primary objective of this study is to evaluate the safety of hydrocodone extended-release tablets when used over a 12-month period in patients with chronic pain, as assessed by adverse events, clinical laboratory results, vital signs measurements, electrocardiogram results, physical examination findings, pure tone audiometry, and concomitant medication usage.

DETAILED DESCRIPTION:
This was a Phase 3, open-label, nonrandomized study that consisted of a screening period, an open label titration period, and a 52 week, long term, open-label treatment period in patients with chronic pain. Patients were eligible to participate in this study if they had completed study C33237/3079 (NCT01240863) (these patients are hereafter referred to as rollover patients) or if they had not participated in study 3079 (these patients are hereafter referred to as either new opioid naïve or new opioid experienced patients).

ELIGIBILITY:
Inclusion Criteria:

* The patient must be willing and able to successfully self-administer the study drug, comply with study restrictions, and return to the clinic for scheduled study visits as specified in this protocol.
* The patient has either completed Cephalon study 3079 or has chronic pain of at least 3 months duration prior to entering this study associated with any of the following conditions: diabetic peripheral neuropathy, postherpetic neuralgia, traumatic injury, complex regional pain syndrome, back pain, neck pain, osteoarthritis, or rheumatoid arthritis. Patients with other painful conditions may qualify for the study with permission from the Cephalon medical monitor or designee.
* Those patients who completed the 12-week, double-blind, placebo-controlled, randomized study (study 3079) and are willing to re-titrate study drug to an effective dose of hydrocodone extended-release tablets are eligible to enter this study.
* The patient is able to speak English, willing to provide written informed consent, and sign a written opioid agreement, to participate in this study.
* The patient is 18 through 80 years of age (inclusive) at the time of entering this or the previous study (study 3079).
* Women of childbearing potential (not surgically sterile or 2 years postmenopausal), must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after participation in the study, and have a negative pregnancy test at screening.

Exclusion Criteria:

* Patients who were enrolled in study 3079 but did not complete the 12-week, double-blind, placebo-controlled, randomized study may not be enrolled into this study.
* The patient has known or suspected hypersensitivities, allergies, or other contraindications to the study drug or its excipients.
* The patient has a recent history (within 5 years) or current evidence of alcohol or other substance abuse.
* The patient has a medical or psychiatric condition/disease that, in the opinion of the investigator, would compromise collected data.
* The patient is taking a total (i.e., including around-the clock [ATC] and rescue medications) of more than 135 mg/day of oxycodone or equivalent for 14 days prior to screening.
* The patient has a history of suicidality.
* The patient has a diagnosis of chronic headache or migraine as the primary painful condition under study.
* The patient is expected to have surgery during the study and it is anticipated that the surgery will alleviate the patient's pain.
* The patient is pregnant or lactating.
* The patient has active malignancy.
* The patient has human immunodeficiency virus (HIV).
* In the judgment of the investigator, the patient has any clinically significant deviation from normal in the physical examination and/or clinical laboratory test values.
* The patient has cardiopulmonary disease that would, in the opinion of the investigator, significantly increase the risk of treatment with potent synthetic opioids.
* The patient has participated in a study involving an investigational drug in the previous 30 days (excluding those who participated in study 3079).
* The patient has received a monoamine oxidase inhibitor (MAOI) within 14 days before the first treatment with study drug.
* The patient has any other medical condition or is receiving concomitant medication/therapy (e.g., regional nerve block) that would, in the opinion of the investigator, compromise the patient's safety or compliance with the study protocol, or compromise collected data.
* The patient is involved in active litigation in regard to the chronic pain currently being treated.
* The patient has a positive urine drug screen (UDS) for an illicit substance or medication not prescribed by the physician currently treating the chronic pain.
* The investigator feels that the patient is not suitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, MD, Study Director — Cephalon
Locations (54):
- United States (54):
  - Horizon Research Group, LLC, Mobile, Alabama
  - Physician Alliance Research Center, Anaheim, California
  - Adam D. Karns, MD, Beverly Hills, California
  - Associated Pharmaceutical Research Center, Inc., Buena Park, California
  - Providence Clinical Research, Burbank, California
  - Research Center of Fresno, Inc., Fresno, California
  - Pacific Coast Pain Management Center, Laguna Hills, California
  - South Orange County Surgical Medical Group, Laguna Hills, California
  - Accelovance, Inc., San Diego, California
  - Bayview Research Group, LLC, Valley Village, California
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Compass Research, LLC, Orlando, Florida
  - Sarasota Pain Medicine Research LLC, Sarasota, Florida
  - Gold Coast Research LLC, Weston, Florida
  - Drug Studies America, Marietta, Georgia
  - Georgia Institute for Clinical Research, LLC, Marietta, Georgia
  - Taylor Research, LLC, Marietta, Georgia
  - Better Health Clinical Research, Inc., Newnan, Georgia
  - Millennium Pain Center, Bloomington, Illinois
  - Rehabilitation Associates of Indiana, Indianapolis, Indiana
  - International Clinical Research, Inc., Overland Park, Kansas
  - Community Research, Crestview Hills, Kentucky
  - Willis Knighton River Cities Clinical Research Center, Shreveport, Louisiana
  - MidAtlantic Pain Medicine Center, Pikesville, Maryland
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - HealthCare Research, Florissant, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Meridian Clinical Research, Omaha, Nebraska
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Advanced Pain Consultants, Voorhees Township, New Jersey
  - Upstate Clinical Research Associates, Williamsville, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - Columbus Clinical Research, Columbus, Ohio
  - SP Research, Oklahoma City, Oklahoma
  - Pain Research of Oregon, Eugene, Oregon
  - Summit Research Network Inc., Portland, Oregon
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - AMH Feasterville Family Health Care Center, Feasterville-Trevose, Pennsylvania
  - Tipton Medical and Diagnostic Center, Tipton, Pennsylvania
  - Clinical Research Center of Reading, LLP, West Reading, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Greenville Pharmaceutical Research, Greenville, South Carolina
  - Trident Institute of Medical Research, LLC, North Charleston, South Carolina
  - S. Carolina Pharmaceutical Research, Spartanburg, South Carolina
  - KRK Medical Research, Dallas, Texas
  - Radiant Research, Dallas, Texas
  - Renaissance Clinical Research & Hypertension of Texas, PLLC, Dallas, Texas
  - Medstar Clinical Research, Houston, Texas
  - Benchmark Research, San Angelo, Texas
  - DCT-Sugarland, LLC dba Discovery Clinical Trials, Sugar Land, Texas
  - Hillcrest Family Health Centers, Waco, Texas
  - Aspen Clinical Research, LLC, Orem, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 365 patients with chronic pain were screened for enrollment into this study: 25 patients were excluded on the basis of exclusion criteria, 6 withdrew consent, 2 were lost to follow up before the baseline visit, 1 patient did not meet an inclusion criteria, and 1 patient had an opioid violation because of self increasing analgesic medication.
Pre-assignment Details: 330 enrolled patients came from 61 centers in the US: 166 rolled-over from study 3079, 52 were new opioid-naïve participants and 112 were new opioid-experienced participants. One enrolled patient was withdrawn before taking any study drug.
Groups:
- Hydrocodone ER: Participants were titrated (or re-titrated for roll-over participants) at escalating dosages of hydrocodone ER tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours until deemed successful for managing their pain during the open-label titration period. Once a successful dose was identified, participants entered the 52 week open-label treatment period in which hydrocodone ER was administered at the successful dose (15, 30, 45, 60, or 90 mg) every 12 hours.
Period: Open-label Titration Period
Arm/Group | Hydrocodone ER
Started | 330
Safety Analysis Set | 329
Achieved Stable Pain Relief | 294
Completed | 291
Not Completed | 39
Not completed — Enrolled but not treated | 1
Not completed — Adverse Event | 23
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 5
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 2
Not completed — Noncompliance with study drug admin | 1
Not completed — Noncompliance with study procedures | 2
Not completed — Starting physical therapy | 1
Period: Open-label Treatment Period
Arm/Group | Hydrocodone ER
Started | 291
Completed | 189
Not Completed | 102
Not completed — Adverse Event | 39
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 19
Not completed — Protocol Violation | 15
Not completed — Lost to Follow-up | 7
Not completed — Noncompliance with study drug admin | 7
Not completed — Noncompliance with study procedures | 6
Not completed — Moved out of area | 2
Not completed — Negative urine drug screen when on treat | 1
Not completed — "Out of window" | 1
Not completed — Starting physical therapy | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: Enrolled patients
Groups:
- Hydrocodone ER: Participants were titrated (or re-titrated for roll-over participants) at escalating dosages of hydrocodone ER tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours until deemed successful for managing their pain during the open-label titration period. Once a successful dose was identified, participants entered the 52 week open-label treatment period in which hydrocodone ER was administered at th3 successful dose (15, 30, 45, 60, or 90 mg) every 12 hours.
Arm/Group | Hydrocodone ER
Number analyzed (Participants) | 330
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197
  Male | 133
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 260
  Black | 66
  Asian | 2
  Pacific Islander | 1
  Other | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Non-Hispanic and non-Latino | 319
  Unknown | 1
Weight [Mean (Standard Deviation); unit: kg] — Population: one participant data was missing the value
  kg
    number analyzed (Participants) | 329
    (all) | 95.6 (23.97)
Height [Mean (Standard Deviation); unit: cm] — Population: one participant data was missing the value
  cm
    number analyzed (Participants) | 329
    (all) | 169.7 (10.57)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: one participant data was missing the value
  kg/m^2
    number analyzed (Participants) | 329
    (all) | 33.1 (7.38)
Type of Pain [Count of Participants; unit: Participants]
  Low back pain | 113
  Back pain | 103
  Osteoarthritis | 82
  Diabetic peripheral neuropathy | 12
  Postherpetic neuralgia | 0
  Traumatic injury | 3
  Neck pain | 10
  Complex regional pain syndrome | 3
  Rheumatoid arthritis | 2
  Other | 2
Duration Since Diagnosis [Mean (Standard Deviation); unit: years] | 12.3 (9.54)
Duration on Opioid Therapy [Mean (Standard Deviation); unit: years] | 4.4 (5.27)

OUTCOME MEASURES:

1. Primary Outcome: Participants With Adverse Experiences
Description: An adverse event (AE) was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 of open-label titration period - Week 52 of the open-label treatment period
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Groups:
- New Opioid Naïve Subpopulation: The subpopulation of participants who enrolled in this study without previous participation in study C33237/3079 (NCT01240863) and were categorized as opioid naïve (ie, those who were taking less than 10 mg/day of oxycodone or equivalent for the 14 days immediately before screening).
- New Opioid Experienced Subpopulation: The subpopulation of participants who enrolled in this study without previous participation in study C33237/3079 (NCT01240863) and were categorized as opioid experienced (ie, those who were taking 10 mg/day or more of oxycodone or equivalent, but not more than 135 mg/day, including around-the-clock medication and rescue medications, for the 14 days immediately before screening).
- Rollover Subpopulation: The subpopulation of participants who completed study C33237/3079 (NCT01240863) and 'rolled over' to participate in this study.
- Total Hydrocodone ER: Participants were titrated (or re-titrated for roll-over participants) at escalating dosages of hydrocodone ER tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours until deemed successful for managing their pain during the open-label titration period. Once a successful dose was identified, participants entered the 52 week open-label treatment period in which hydrocodone ER was administered at a successful dose (15, 30, 45, 60, or 90 mg) every 12 hours.
Arm/Group | New Opioid Naïve Subpopulation | New Opioid Experienced Subpopulation | Rollover Subpopulation | Total Hydrocodone ER
Number analyzed (Participants) | 52 | 112 | 165 | 329
Participants
  Any adverse event | 51 | 98 | 135 | 284
  Treatment-related adverse event | 41 | 69 | 63 | 173
  Death | 0 | 1 | 1 | 2
  Serious adverse event | 4 | 16 | 7 | 27
  Withdrawals from treatment due to adverse event | 18 | 24 | 20 | 62

2. Primary Outcome: Participants With Potentially Clinically Significant (PCS) Abnormal Laboratory Values During the Open-Label Treatment Period by Participant Status
Description: Data represents participants with PCS abnormal serum chemistry, hematology and urinalysis values.
  Significance criteria:
  * alanine aminotransferase (ALT): >=3 times the upper limit of normal (ULN). Normal range is 6-43 U/L
  * aspartate aminotransferase (AST): >=3 times ULN. Normal range is 9-36 U/L
  * blood urea nitrogen (BUN): >=10.71 mmol/L
  * creatinine: >=177 μmol/L
  * uric acid: M>=625, F>=506 μmol/L
  * white blood cell count: <=3.0*10^9/L
  * hemoglobin: M<=115, F<=95 g/dL
  * hematocrit: M<0.37, F<0.32 L/L
  * urine blood (hemoglobin): >=2 unit increase from baseline
  * urine glucose: >=2 unit increase from baseline
Time Frame: Day 1 - Week 52 of the open-label treatment period
Population: Posttitration Safety Analysis set. The posttitration safety analysis set included all patients who successfully completed the open label titration period and received 1 or more doses of study drug treatment in the open label treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | New Opioid Naïve Subpopulation | New Opioid Experienced Subpopulation | Rollover Subpopulation | Total Hydrocodone ER
Number analyzed (Participants) | 42 | 92 | 157 | 291
Participants
  ALT: number analyzed (Participants) | 41 | 89 | 152 | 282
  ALT | 0 | 2 | 1 | 3
  AST: number analyzed (Participants) | 40 | 89 | 152 | 281
  AST | 0 | 2 | 0 | 2
  BUN: number analyzed (Participants) | 41 | 90 | 152 | 283
  BUN | 0 | 3 | 5 | 8
  Creatinine: number analyzed (Participants) | 41 | 90 | 152 | 283
  Creatinine | 0 | 1 | 1 | 2
  Uric acid: number analyzed (Participants) | 41 | 90 | 152 | 283
  Uric acid | 1 | 4 | 3 | 8
  White blood cell count: number analyzed (Participants) | 41 | 90 | 152 | 283
  White blood cell count | 0 | 1 | 0 | 1
  Hemoglobin: number analyzed (Participants) | 41 | 90 | 152 | 283
  Hemoglobin | 1 | 3 | 3 | 7
  Hematocrit: number analyzed (Participants) | 41 | 90 | 152 | 283
  Hematocrit | 2 | 6 | 6 | 14
  Urine blood: number analyzed (Participants) | 41 | 89 | 151 | 281
  Urine blood | 1 | 4 | 2 | 7
  Urine glucose: number analyzed (Participants) | 41 | 89 | 151 | 281
  Urine glucose | 2 | 2 | 5 | 9

3. Primary Outcome: Participants With Potentially Clinically Significant Abnormal Vital Signs Values by Participant Status
Description: Data represents participants with potentially clinically significant (PCS) vital sign values.
  Significance criteria
  * Pulse - high: >=120 and increase of >= 15 beats/minute from baseline
  * Pulse - low: <=50 and decrease of >=15 beats/minute
  * Systolic blood pressure - high: >=180 and increase >=20 mmHg
  * Systolic blood pressure - low: <=90 and decrease >=20 mmHg
  * Diastolic blood pressure - high: >=105 and increase of >=15 mmHg
  * Diastolic blood pressure - low: <=50 and decrease of >=15 mmHg
Time Frame: Day 1 of open-label titration period - Week 52 of the open-label treatment period
Population: Safety analysis set. One rollover participant did not have vital signs values.
Measure: Count of Participants; unit: Participants
Arm/Group | New Opioid Naïve Subpopulation | New Opioid Experienced Subpopulation | Rollover Subpopulation | Total Hydrocodone ER
Number analyzed (Participants) | 52 | 112 | 164 | 328
Participants
  Pulse - high | 0 | 2 | 0 | 2
  Pulse - low | 1 | 0 | 5 | 6
  Systolic blood pressure - high | 1 | 0 | 2 | 3
  Systolic blood pressure - low | 0 | 4 | 7 | 11
  Diastolic blood pressure - high | 3 | 0 | 3 | 6
  Diastolic blood pressure - low | 1 | 2 | 3 | 6

4. Primary Outcome: Shifts in Electrocardiogram (ECG) Findings From Baseline to Overall Study by Participant Status
Description: A 12-lead ECG was conducted at screening, week 24, and week 52 or at the last postbaseline observation. For rollover participants, the ECG performed at the final visit of study 3079 served as the 1st ECG in study 3080. A qualified physician was responsible for interpreting the ECG. Any ECG finding that was judged by the investigator as a clinically meaningful change (worsening) compared with baseline was considered an adverse event.
  For overall results, the worst postbaseline finding for the participant was summarized.
  Results below are formatted as Baseline ECG result - Overall ECG result.
Time Frame: Baseline for new participants was between Day -7 and -14 (the study 3080 screening visit); baseline for rollover participants was the last ECG in study 3079. During study ECGs were performed on weeks 24 and 52 of the open-label treatment period
Population: Post-titration Safety analysis set. Only those participants with both baseline and visit electrocardiogram findings were summarized.
Measure: Count of Participants; unit: Participants
Arm/Group | New Opioid Naïve Subpopulation | New Opioid Experienced Subpopulation | Rollover Subpopulation | Total Hydrocodone ER
Number analyzed (Participants) | 41 | 89 | 150 | 280
Participants
  Normal baseline - Normal overall | 18 | 33 | 43 | 94
  Normal baseline - Abnormal overall | 8 | 17 | 35 | 60
  Abnormal baseline - Normal overall | 0 | 7 | 18 | 25
  Abnormal baseline - Abnormal overall | 15 | 32 | 54 | 101

5. Primary Outcome: Participants With Clinically Significant (CS) Hearing Changes From Baseline in Pure Tone Audiometry Test Results by Patient Status
Description: Pure tone audiometry was performed by trained personnel. During the test, the patient wore headphones and was seated in a quiet room; trained personnel manipulated the audiometry equipment to test the patient's hearing. For serial audiograms, the criteria for a clinically significant (CS) hearing change were based on the guidance from the American Speech-Language Hearing Association (ASHA) 1994 (Konrad-Martin et al 2005). These criteria included the following: greater than 20 decibels (dB) pure tone threshold shift at 1 frequency; greater than 10 dB shift at 2 consecutive test frequencies; or threshold response shifting to "no response" at 3 consecutive test frequencies.
Time Frame: Baseline for new participants was between Day -7 and -14 (study 3080 screening visit); baseline for rollover participants was the baseline test in study 3079. During study covers both open-label titration and 52-week treatment periods
Population: Safety analysis set. The endpoint value is from the post-titration safety set (n=42, 92, 157, 291)
Measure: Count of Participants; unit: Participants
Arm/Group | New Opioid Naïve Subpopulation | New Opioid Experienced Subpopulation | Rollover Subpopulation | Total Hydrocodone ER
Number analyzed (Participants) | 52 | 112 | 165 | 329
Participants
  >=1 CS value during study | 10 | 30 | 36 | 76
  >=1 CS value during open-label titration period | 4 | 14 | 4 | 22
  >=1 CS value at endpoint | 2 | 8 | 13 | 23

6. Secondary Outcome: Participant Global Assessment (PGA) of the Method of Pain Control by Participant Status
Description: The PGA of the method of pain control consisted of a asking patients a single question to assess their method of pain control during the previous 24 hours as either poor, fair, good, or excellent (Rothman et al 2009).
Time Frame: Baseline for new participants was Day 1, i.e. the first day of open-label titration. Baseline for rollover participants was the baseline in study 3079. Week 4 (end of titration, start of open-label treatment), Week 52, last visit up to Week 52
Population: Full analysis set included all patients in the safety analysis set who had at least 1 postbaseline efficacy assessment. Participants contributing to each time point are listed in the time point label.
Measure: Count of Participants; unit: Participants
Arm/Group | New Opioid Naïve Subpopulation | New Opioid Experienced Subpopulation | Rollover Subpopulation | Total Hydrocodone ER
Number analyzed (Participants) | 42 | 92 | 157 | 291
Participants
  Baseline: Poor: number analyzed (Participants) | 34 | 86 | 152 | 272
  Baseline: Poor | 18 | 10 | 49 | 77
  Baseline: Fair: number analyzed (Participants) | 34 | 86 | 152 | 272
  Baseline: Fair | 14 | 55 | 71 | 140
  Baseline: Good | 1 | 18 | 29 | 48
  Baseline: Excellent | 1 | 3 | 3 | 7
  Week 4: Poor: number analyzed (Participants) | 40 | 87 | 150 | 277
  Week 4: Poor | 2 | 1 | 2 | 5
  Week 4: Fair: number analyzed (Participants) | 40 | 87 | 150 | 277
  Week 4: Fair | 5 | 17 | 27 | 49
  Week 4: Good: number analyzed (Participants) | 40 | 87 | 150 | 277
  Week 4: Good | 20 | 54 | 94 | 168
  Week 4: Excellent: number analyzed (Participants) | 40 | 87 | 150 | 277
  Week 4: Excellent | 13 | 15 | 27 | 55
  Week 52: Poor: number analyzed (Participants) | 28 | 57 | 103 | 188
  Week 52: Poor | 0 | 2 | 2 | 4
  Week 52: Fair: number analyzed (Participants) | 28 | 57 | 103 | 188
  Week 52: Fair | 3 | 9 | 18 | 30
  Week 52: Good: number analyzed (Participants) | 28 | 57 | 103 | 188
  Week 52: Good | 17 | 36 | 62 | 115
  Week 52: Excellent: number analyzed (Participants) | 28 | 57 | 103 | 188
  Week 52: Excellent | 8 | 10 | 21 | 39
  Endpoint: Poor | 3 | 6 | 8 | 17
  Endpoint: Fair (n=42, 92, 157, 291) | 7 | 21 | 27 | 55
  Endpoint: Good | 21 | 52 | 93 | 166
  Endpoint: Excellent | 11 | 13 | 29 | 53

7. Secondary Outcome: Participants by Risk Category for Aberrant Drug Misuse Based on the Total Score in the Screener and Opioid Assessment for Patients With Pain - Revised (SOAPP-R)
Description: SOAPP-R is a clinician-rated scale used to assess each patient's risk of developing aberrant drug use behaviors while on long term opioid therapy. SOAPP-R consists of 24 questions that address 8 concepts: substance abuse history, medication related behaviors, antisocial behaviors/history, psychosocial problems, psychiatric history, physician patient relationship factors, emotional attachment to pain medications, and personal care and lifestyle issues (Butler et al 2008). Each question is answered using a 5 point Likert-like scale, with 0=never, 1=seldom, 2=sometimes, 3=often, and 4=very often for a total range of 0-96. The higher the overall score, the greater the probability the patient is at risk for displaying aberrant behaviors consistent with drug use.
  An overall score of 18 or higher is considered positive for predicting aberrant drug related behavior, therefore the reported risk categories are
  * <18 and
  * <=18. Results indicate timeframe followed by risk cat
Time Frame: End of Open-label Titration Period. Weeks 4 and 24 of the Open-label Treatment Period
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | New Opioid Naïve Subpopulation | New Opioid Experienced Subpopulation | Rollover Subpopulation | Total Hydrocodone ER
Number analyzed (Participants) | 52 | 112 | 165 | 329
Participants
  End of Open-Label Titration: >=18 | 0 | 0 | 0 | 0
  End of Open-Label Titration: <18 | 0 | 0 | 2 | 2
  Week 4: >=18 | 1 | 12 | 3 | 16
  Week 4: <18 | 39 | 73 | 134 | 246
  Week 24: >=18 | 0 | 0 | 0 | 0
  Week 24: <18 | 0 | 0 | 1 | 1

8. Secondary Outcome: Addiction Behavior Checklist (ABC) Total Scores During Both the Open-Label Titration and Open-Label Treatment Periods by Participant Status
Description: The ABC was a clinician rated scale that consisted of a brief (21 item) questionnaire designed to track behaviors characteristic of addiction related to prescription opioid medications in chronic pain populations. Items were focused on observable behaviors noted both during and between clinic visits. Each affirmative response was counted as 1 point, and points were added to calculate the total score. All but 1 of the 21 items (the provider's impression) was used in calculating the total score, consequently resulting in scores ranging from 0 to 20 (0=no addiction-related behaviors seen and higher scores indicating an increasing number of addition-related behaviors seen). Participants with a total score of 3 or greater were classified as exhibiting inappropriate opioid use during the study.
Time Frame: Baseline for new participants was Day 1 of open-label titration; rollover participants baseline was in study 3079. End of Open-label Titration: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36 40, 44, 48, 52 and last visit up to week 52
Population: Post-titration Safety Analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | New Opioid Naïve Subpopulation | New Opioid Experienced Subpopulation | Rollover Subpopulation | Total Hydrocodone ER
Number analyzed (Participants) | 42 | 92 | 157 | 291
units on a scale
  Baseline: number analyzed (Participants) | 40 | 90 | 155 | 285
  Baseline | 0.1 (0.40) | 0.1 (0.46) | 0.2 (0.60) | 0.2 (0.53)
  End of Titration: number analyzed (Participants) | 40 | 92 | 157 | 289
  End of Titration | 0.1 (0.22) | 0.0 (0.15) | 0.1 (0.38) | 0.1 (0.31)
  Week 4: number analyzed (Participants) | 40 | 86 | 150 | 276
  Week 4 | 0.2 (0.43) | 0.2 (0.47) | 0.1 (0.39) | 0.1 (0.42)
  Week 8: number analyzed (Participants) | 34 | 76 | 143 | 253
  Week 8 | 0.1 (0.41) | 0.2 (0.42) | 0.1 (0.38) | 0.1 (0.40)
  Week 12: number analyzed (Participants) | 32 | 73 | 137 | 242
  Week 12 | 0.2 (0.51) | 0.2 (0.40) | 0.1 (0.36) | 0.1 (0.39)
  Week 16: number analyzed (Participants) | 31 | 69 | 133 | 233
  Week 16 | 0.1 (0.34) | 0.1 (0.29) | 0.2 (0.56) | 0.1 (0.47)
  Week 20: number analyzed (Participants) | 30 | 67 | 128 | 225
  Week 20 | 0.2 (0.46) | 0.1 (0.24) | 0.2 (0.45) | 0.1 (0.40)
  Week 24: number analyzed (Participants) | 29 | 67 | 123 | 219
  Week 24 | 0.1 (0.26) | 0.1 (0.31) | 0.1 (0.41) | 0.1 (0.36)
  Week 28: number analyzed (Participants) | 29 | 65 | 120 | 214
  Week 28 | 0.1 (0.41) | 0.1 (0.27) | 0.1 (0.42) | 0.1 (0.38)
  Week 32: number analyzed (Participants) | 29 | 63 | 114 | 206
  Week 32 | 0.2 (0.60) | 0.0 (0.25) | 0.1 (0.42) | 0.1 (0.41)
  Week 36: number analyzed (Participants) | 28 | 63 | 109 | 200
  Week 36 | 0.1 (0.59) | 0.1 (0.43) | 0.1 (0.41) | 0.1 (0.44)
  Week 40: number analyzed (Participants) | 28 | 61 | 108 | 197
  Week 40 | 0.1 (0.31) | 0.1 (0.25) | 0.1 (0.46) | 0.1 (0.38)
  Week 44: number analyzed (Participants) | 28 | 59 | 104 | 191
  Week 44 | 0.1 (0.26) | 0.1 (0.31) | 0.1 (0.44) | 0.1 (0.38)
  Week 48: number analyzed (Participants) | 28 | 57 | 104 | 189
  Week 48 | 0.0 (0.19) | 0.0 (0.13) | 0.1 (0.41) | 0.1 (0.32)
  Week 52: number analyzed (Participants) | 28 | 57 | 103 | 188
  Week 52 | 0.1 (0.45) | 0.1 (0.23) | 0.1 (0.41) | 0.1 (0.37)
  Endpoint | 0.2 (0.52) | 0.2 (0.60) | 0.2 (0.59) | 0.2 (0.58)

9. Secondary Outcome: Current Opioid Misuse Measure (COMM) Scores During Both the Open-Label Titration and Open-Label Treatment Periods by Participant Status
Description: The COMM was a clinician-rated scale developed as a brief self-report measure of current aberrant drug-related behavior for patients with chronic pain who were already on long-term opioid therapy. A total score was calculated as the sum of the 17 questions. The total score ranged from 0 to 68. A score of 0 indicates no aberrant drug-related behaviors were seen. Patients with a total score of 9 or greater were classified as exhibiting aberrant drug-related behavior.
Time Frame: Baseline for new participants was Day 1 of open-label titration; rollover participants baseline was in study 3079. End of Open-label Titration Period. Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36 40, 44, 48, 52 and last visit up to week 52
Population: Post titration Safety Analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | New Opioid Naïve Subpopulation | New Opioid Experienced Subpopulation | Rollover Subpopulation | Total Hydrocodone ER
Number analyzed (Participants) | 42 | 92 | 157 | 291
units on a scale
  Baseline: number analyzed (Participants) | 42 | 91 | 157 | 290
  Baseline | 5.1 (5.29) | 5.4 (4.61) | 3.7 (3.70) | 4.4 (4.31)
  End of Titration: number analyzed (Participants) | 42 | 91 | 157 | 290
  End of Titration | 3.8 (3.37) | 4.0 (3.66) | 2.1 (2.74) | 3.0 (3.26)
  Week 4: number analyzed (Participants) | 39 | 86 | 150 | 275
  Week 4 | 3.2 (3.06) | 3.7 (3.70) | 2.3 (2.83) | 2.9 (3.21)
  Week 8: number analyzed (Participants) | 34 | 76 | 143 | 253
  Week 8 | 2.4 (2.44) | 3.9 (4.12) | 2.4 (2.96) | 2.8 (3.36)
  Week 12: number analyzed (Participants) | 32 | 73 | 137 | 242
  Week 12 | 3.1 (3.12) | 4.2 (3.99) | 2.4 (2.71) | 3.1 (3.28)
  Week 16: number analyzed (Participants) | 31 | 69 | 133 | 233
  Week 16 | 2.4 (1.98) | 4.0 (4.84) | 2.3 (2.82) | 2.9 (3.53)
  Week 20: number analyzed (Participants) | 30 | 67 | 128 | 225
  Week 20 | 2.6 (2.49) | 3.5 (3.78) | 2.1 (2.80) | 2.6 (3.13)
  Week 24: number analyzed (Participants) | 29 | 67 | 122 | 218
  Week 24 | 2.6 (2.66) | 3.9 (4.14) | 2.4 (3.04) | 2.9 (3.42)
  Week 28: number analyzed (Participants) | 29 | 65 | 121 | 215
  Week 28 | 2.1 (2.10) | 3.3 (3.66) | 2.3 (2.91) | 2.6 (3.09)
  Week 32: number analyzed (Participants) | 29 | 63 | 114 | 206
  Week 32 | 2.3 (1.84) | 2.8 (3.07) | 2.0 (2.62) | 2.3 (2.69)
  Week 36: number analyzed (Participants) | 28 | 63 | 110 | 201
  Week 36 | 2.9 (2.44) | 3.2 (3.35) | 2.3 (3.30) | 2.7 (3.22)
  Week 40: number analyzed (Participants) | 28 | 61 | 108 | 197
  Week 40 | 2.8 (3.21) | 3.0 (3.20) | 2.1 (2.97) | 2.5 (3.09)
  Week 44: number analyzed (Participants) | 28 | 59 | 105 | 192
  Week 44 | 2.3 (1.90) | 2.7 (2.86) | 2.2 (3.41) | 2.4 (3.06)
  Week 48: number analyzed (Participants) | 28 | 57 | 104 | 189
  Week 48 | 2.4 (2.57) | 3.0 (3.98) | 2.3 (3.19) | 2.5 (3.37)
  Week 52: number analyzed (Participants) | 28 | 57 | 103 | 188
  Week 52 | 2.4 (2.39) | 3.0 (3.30) | 2.3 (3.05) | 2.5 (3.04)
  Endpoint | 3.5 (3.74) | 4.2 (4.41) | 2.5 (3.25) | 3.2 (3.78)

ADVERSE EVENTS:
Time Frame: Day 1 of Open-label Titration period - Week 52 of the Open-label Treatment period
Arm/Group | New Opioid Naïve Subpopulation | New Opioid Experienced Subpopulation | Rollover Subpopulation
Serious Adverse Events (participants affected / at risk) | 4/52 | 16/112 | 7/165
Other Adverse Events (participants affected / at risk) | 47/52 | 83/112 | 109/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | New Opioid Naïve Subpopulation (N=52) | New Opioid Experienced Subpopulation (N=112) | Rollover Subpopulation (N=165)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Listeria sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia cryptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/24 (0) | 1/44 (1) | 0/64 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Impulsive behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | New Opioid Naïve Subpopulation (N=52) | New Opioid Experienced Subpopulation (N=112) | Rollover Subpopulation (N=165)
Constipation (Gastrointestinal disorders) | 19 (22) | 35 (45) | 31 (43)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 8 (9) | 13 (19)
Nausea (Gastrointestinal disorders) | 16 (20) | 18 (25) | 28 (36)
Vomiting (Gastrointestinal disorders) | 8 (9) | 7 (9) | 16 (17)
Fatigue (General disorders) | 3 (3) | 7 (9) | 6 (6)
Oedema peripheral (General disorders) | 3 (3) | 6 (6) | 7 (8)
Bronchitis (Infections and infestations) | 3 (3) | 8 (9) | 6 (8)
Influenza (Infections and infestations) | 5 (7) | 5 (5) | 4 (5)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (5) | 10 (11)
Sinusitis (Infections and infestations) | 0 (0) | 6 (11) | 11 (11)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 6 (7) | 15 (16)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 9 (11) | 6 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 10 (12) | 14 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (9) | 10 (13)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6) | 8 (11)
Dizziness (Nervous system disorders) | 4 (4) | 7 (11) | 6 (7)
Headache (Nervous system disorders) | 8 (11) | 20 (24) | 10 (12)
Mental impairment (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 9 (12) | 15 (16) | 11 (12)
Insomnia (Psychiatric disorders) | 3 (3) | 6 (6) | 7 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (9) | 5 (5)
Hypertension (Vascular disorders) | 4 (4) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.